CLINICAL TRIAL: NCT06295341
Title: Short Stature and Psychological Well-being
Acronym: PSICOSHORT
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C312
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Short Stature; Short; Stature, Psychosocial
Keywords: Short stature; Psychological well-being; Psychological distress; Life quality
MeSH Terms: conditions — Dwarfism; Psychological Well-Being | interventions — Growth Hormone; Single Person

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (3):
- cases - children with familial short stature: - 35 children, aged between 6 and 14 years, of both sexes, with familial short stature (height < 3rd centile according to the Italian reference standards) and their caregivers of reference. Children with familial short stature will be characterized by: short stature in other members of the family group, not necessarily the parents, harmonious appearance, without particular clinical signs and normal pubertal development, parallel growth curve below the 3rd centile, bone age corresponding to chronological age. Children and teenagers with obesity (BMI > 97th centile) will be excluded
- cases - children with normal height: 35 children, aged between 6 and 14 years, of both sexes, with normal height (height > 25th centile) and weight.
- cases - children with growth hormone deficiency: 10 children, aged between 6 and 14 years, of both sexes, affected by isolated GH deficiency according to the criteria established by AIFA note 39 for this pathology (short stature: ≤ -3 SD or ≤ -2 SD and growth velocity/year ≤ -1.0 SD for age and sex evaluated at least 6 months apart and peak GH at two different pharmacological stimulus tests < 8 ng/ml). The exclusion criterion from the present study (and from treatment with rhGH) will be the presence of organic pathologies at the hypothalamic-pituitary level (assessed by performing brain MRI).
  Children with GH deficiency are evaluated in baseline conditions and after 6 months of therapy with recombinant DNA GH (at a dose of 0.025-0.035 mg/kg of body weight per day (or 0.7-1.0 mg/m2 of body surface area per day).
  Interventions: Drug: Recombinant human growth hormone (only for children with growth hormone deficiency)

INTERVENTIONS:
Drug: Recombinant human growth hormone (only for children with growth hormone deficiency) — 6 months of therapy with recombinant DNA GH (at a dose of 0.025-0.035 mg/kg of body weight per day (or 0.7-1.0 mg/m2 of body surface area per day).
  Groups: cases - children with growth hormone deficiency

SUMMARY:
The first aim of the present study is to evaluate the psychological impact of the condition of short stature (family) in a sample of Italian children, comparing them with subjects of normal stature, measuring their levels of psychological well-being, psychological distress, quality of health-related life and any behavioral issues. The secondary objective is to study the psychological impact evaluated with the tests described below (see methods section) in children with GH deficiency and the effects of replacement therapy (6 months) with GH from recombinant DNA.

DETAILED DESCRIPTION:
The observational study carried out at the Centre for growth and pubertal Disorders, Istituto Auxologico Italiano, IRCCS, Milan, consists of two sub-projects that involve the recruitment of:

* 70 children, aged between 6 and 14 years, of both sexes: 35 with familiar short stature (height < 3rd centile according to the Italian reference standards) and 35 with normal height (height > 25th centile), of normal weight, and their caregivers of reference. Children with familial short stature will be characterized by: short stature in other members of the family group, not necessarily the parents, harmonious appearance, without particular clinical signs and normal pubertal development, parallel growth curve below the 3rd centile, bone age corresponding to chronological age. Children and teenagers with obesity (BMI > 97th centile) will be excluded
* 10 children, aged between 6 and 14 years, of both sexes, affected by isolated GH deficiency according to the criteria established by AIFA note 39 for this pathology (short stature: ≤ -3 SD or ≤ -2 SD and growth velocity/year ≤ -1.0 SD for age and sex evaluated at least 6 months apart and peak GH at two different pharmacological stimulus tests < 8 ng/ml). The exclusion criterion from the present study (and from treatment with rhGH) will be the presence of organic pathologies at the hypothalamic-pituitary level (assessed by performing brain MRI).

Children with GH deficiency will be evaluated in baseline conditions and after 6 months of therapy with recombinant DNA GH (at a dose of 0.025-0.035 mg/kg of body weight per day (or 0.7-1.0 mg/m2 of body surface area per day).

The following variables will be investigated in the recruited subjects of the two subgroups:

* socio-demographic conditions (gender, age, provenance, level of education, family composition)
* psychological well-being through the Psychological Well-Being Scales (PWB), a self-administered questionnaire consisting of 18 items that investigates the degree of psychological well-being by exploring six dimensions: self-acceptance, positive relationships with others, autonomy, environmental control, personal growth, and purpose of life. The questionnaire consists of 18 items on a 4-step Likert scale.
* psychological distress through the Depression Anxiety Stress Scale (DASS-21), a 21-item self-report tool that measures various negative internal states: depression, anxiety, and stress.
* quality of life through the Quality of Life in Short Stature Youth (QoLISSY), a 50-item domain-specific questionnaire that measures health-related quality of life in children with short stature.
* skills and problems through the Strengths and Difficulties Questionnaire (SDQ), a questionnaire made up of 25 items able to assess emotional symptoms, behavioral problems, hyperactivity/inattention, problematic relationships with peers, and prosocial behavior.
* behavioral problems through the Child Behaviour Checklist for Children (CBCL), a questionnaire to be administered to parents or caregivers of children who are able to detect any behavioral problems. The instrument consists of 113 items that investigate three general scales: total problems, internalizing problems, and externalizing problems and 8 syndromic scales: social withdrawal, somatic complaints, anxiety, depression, social problems, thinking problems, attention problems, antisocial behavior, and aggressive behavior).

ELIGIBILITY:
Inclusion Criteria: age between 6 and 14 years, of both sexes

* 35 with familiar short stature (height < 3rd centile according to the Italian reference standards) and their caregivers of reference. Children with familial short stature are characterized by: short stature in other members of the family group, not necessarily the parents, harmonious appearance, without particular clinical signs and normal pubertal development, parallel growth curve below the 3rd centile, bone age corresponding to chronological age.
* 35 with normal height (height > 25th centile), aged between 6 and 14 years, of normal weight, and their caregivers of reference
* 10 children, aged between 6 and 14 years, of both sexes, affected by isolated GH deficiency according to the criteria established by AIFA note 39 for this pathology (short stature: ≤ -3 SD or ≤ -2 SD and growth velocity/year ≤ -1.0 SD for age and sex evaluated at least 6 months apart and peak GH at two different pharmacological stimulus tests < 8 ng/ml) and their caregivers of reference

Exclusion Criteria:

* children and teenagers with obesity (BMI > 97th centile) are excluded (for the subgroups with familiar short stature or normal height
* children and teenagers with the presence of organic pathologies at the hypothalamic-pituitary level (assessed by performing brain MRI) (for the subgroup with growth hormone deficiency)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 35 children with familiar short stature, 35 with normal height (height > 25th centile), and 10 with growth hormone deficiency and their caregivers of reference (see above the description of the diagnostic criteria).
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Psychological well-being through the Psychological Well-Being Scales (PWB) | Baseline for the three groups; baseline and after 6 months for children with growth hormone deficiency
  A self-administered questionnaire consisting of 18 items that investigates the degree of psychological well-being by exploring six dimensions: self-acceptance, positive relationships with others, autonomy, environmental control, personal growth, and purpose of life. The questionnaire consists of 18 items on a 4-step Likert scale.
Psychological distress through the Depression Anxiety Stress Scale (DASS-21) | Baseline for the three groups; baseline and after 6 months for children with growth hormone deficiency
  A 21-item self-report tool that measures various negative internal states: depression, anxiety, and stress.
Quality of life through the Quality of Life in Short Stature Youth (QoLISSY), | Baseline for the three groups; baseline and after 6 months for children with growth hormone deficiency
  A 50-item domain-specific questionnaire that measures health-related quality of life in children with short stature.
Skills and problems through the Strengths and Difficulties Questionnaire (SDQ) | Baseline for the three groups; baseline and after 6 months for children with growth hormone deficiency
  A questionnaire made up of 25 items able to assess emotional symptoms, behavioral problems, hyperactivity/inattention, problematic relationships with peers, and prosocial behavior.

SECONDARY OUTCOMES:
Behavioral problems through the Child Behaviour Checklist for Children (CBCL) | Baseline for the three groups; baseline and after 6 months for the parents of children with growth hormone deficiency
  A questionnaire to be administered to parents or caregivers of children to detect any behavioral problems in their children. The instrument consists of 113 items that investigate three general scales: total problems, internalizing problems, and externalizing problems and 8 syndromic scales: social withdrawal, somatic complaints, anxiety, depression, social problems, thinking problems, attention problems, antisocial behavior, and aggressive behavior).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy